CLINICAL TRIAL: NCT01736891
Title: Evaluation for the Efficacy,Tolerability,and Safety of Rasagiline in Levodopa-treated PD Patients With Motor Fluctuations: A Multicenter, Double Blind, Randomized, Placebo-Controlled Group Study (China)
Brief Title: Clinical Trial of Rasagiline in Levodopa-Treated Parkinson's Disease Patients With Motor Fluctuations
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chongqing Fortune Pharmaceutical Co., Ltd. (Industry)
Collaborators: Beijing Bionovo Medicine Development Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RLPDMF2010L03416
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2012-11

CONDITIONS: Parkinson´s Disease
Keywords: Motor fluctuations; Parkinson´s Disease; Rasagiline
MeSH Terms: conditions — Parkinson Disease | interventions — rasagiline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rasagiline (Experimental): Rasagiline 0.5 mg by mouth every day for 2 weeks, then 1 mg by mouth every day for 12 weeks, then switch to 0.5mg by mouth every day for remainder of the study (approximately 16 weeks total)
  Interventions: Drug: Rasagiline
- Placebo (Placebo Comparator): placebo 0.5 mg by mouth every day for two weeks, then 1 mg by mouth every day for 12 weeks, then switch to 0.5mg by mouth every day for remainder of the study (approximately 16 weeks total)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rasagiline — Tablets, qd
  Other Names: Azilect
  Arms: Rasagiline
Drug: Placebo — Tablets, qd
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the efficacy, tolerability, and safety of rasagiline compared to placebo in PD patients with motor fluctuations on levodopa therapy.

DETAILED DESCRIPTION:
Levodopa has been the mainstay therapy for PD for decades, and it is considered to be one of the most effective medications for relief of the symptoms of PD. However, within few months to few years the majority of levodopa-treated patients notice a decline in the duration of benefit of each dose and develop motor-complications. A major problem is the appearance of fluctuations in mobility, cycles of ON and OFF periods. The administration of rasagiline, a MAO-B inhibitor, can slow the elimination of the endogenous dopamine supplies or the dopamine produced from the exogenous levodopa therapy and may therefore improve ON-OFF fluctuations.

The objective of this study is to evaluate the efficacy, tolerability, and safety of rasagiline compared to placebo in PD patients with motor fluctuations on levodopa therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic PD
* Patients receiving at least 300 mg daily doses of levodopa and not less than 8 daily doses of levodopa with the stable dose
* Patient with a Modified Hoehn and Yahr stage between 2 to 4 in the OFF state
* Patient with motor fluctuations averaging at least 2 hour daily in the OFF state
* Patients who have demonstrated the ability to keep accurate 24-hour diaries

Exclusion Criteria:

* Patients with Parkinsonian syndrome induced by medicine, metabolic disease, Encephalitis and central nervous system degenerative diseases or Disease of basal ganglia
* Patients with severe cognitive impairment judged by a Mini Mental State Examination
* Patients with a clinically significant psychiatric illness
* Patients with Hamilton Depression Rating Scale (HAMD): total score ≤10
* Patients with a clinically significant or unstable medical or surgical condition which would preclude safe and complete study participation
* Patients with a clinically significant or unstable vascular disease
* Patients with severe disabling dyskinesias Other inclusion and exclusion criteria may apply

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2011-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Efficacy of rasagiline vs placebo as assessed by the change from baseline to week 14 in mean total daily OFF time measured by patients' home diaries in levodopa-treated PD patients with motor fluctuations. | 0, 14 weeks

SECONDARY OUTCOMES:
Change from baseline to week 6/10/16 in mean total daily OFF time measured by patients' home diaries. | 0, 6, 10, 16 weeks
Change from baseline to week 6/14/16 in mean total daily ON time measured by patients' home diaries. | 0, 6, 14, 16 weeks
Change from baseline to week 6/14/16 on Unified Parkinson's Disease Rating Scale (UPDRS) Ⅱ- Ⅵ Activities of Daily Living. | 0, 6, 14, 16 weeks
Change from baseline to week 6/10/14/16 in mean total daily ON time measured by patients' home diaries. | 0, 6, 10, 14, 16 weeks
Analysis of the changing rate of the UPDRSⅡ -Ⅵ after treatment of week 6/14/16. | 0, 6, 14, 16 weeks
The rate of patients whose Levodopa dose is adjusted after 6/14/16 weeks of treatment. | 0, 2, 6, 14, 16 weeks
BP、 temperature、 breath and heart rate after 5 minutes of stasis. | -2, 0, 2, 6, 10, 14, 16 weeks
Physical examination. | -2, 16 weeks
Adverse Events: the occurrence of melanoma. | 0, 2, 6, 10, 14, 16 weeks
Grade of UPDRS I | 0, 6, 14, 16 weeks
Blood routine、 urine routine、 ALT、 AST、 TBiL、 γ-GTP、 ALP、 BUN、 Cr、 ECG. | 0, 6, 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gang Zhao, Principal Investigator — The First Affiliated Hospital of the Fourth Military Medical University
Locations (8):
- China (8):
  - CN002, Chengdu
  - CN005, Chenzhou
  - CN007, Chongqing
  - CN003, Guilin
  - CN004, Lanzhou
  - CN006, Luzhou
  - CN008, Nanjing
  - CN001, Xi'an